CLINICAL TRIAL: NCT00646906
Title: A Randomized, Double-Blind, Crossover Study to Evaluate the Mechanism of Action of Acetaminophen
Brief Title: Mechanisms of Action of Acetaminophen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 708270
Record Dates: First submitted 2008-03-26; First posted 2008-03-31 (Estimated); Results first posted 2019-12-03 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Myocardial Infarction; Arthritis
Keywords: acetaminophen; low dose aspirin; cyclooxygenase; prostaglandin; drug interaction; platelet inhibition; urinary prostaglandin metabolites; oxidant stress; smoking
MeSH Terms: conditions — Myocardial Infarction; Arthritis; Smoking | interventions — Acetaminophen; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Phase 1a: Acetaminophen 1000mg / aspirin (Experimental): All subjects in this arm (smokers (n=8) and non-smokers (n=8) will receive 81 mg aspirin at approximately 8 am followed by 1000 mg acetaminophen at approximately 10 am during one crossover period (see "Crossover period: Aspirin first" intervention). During the other crossover period, beginning after a 2 week washout, the order will be reversed and the subjects will receive 1000 mg acetaminophen at 8 am followed by 81 mg aspirin at 10 am (see "Crossover Period: Aspirin last" intervention). The occurrence of the two crossover periods will be randomized by order. Smokers and non-smokers will be matched for age and gender.
  Interventions: Drug: Aspirin First; Drug: Aspirin Last
- Phase 1a: Acetaminophen 2000mg / aspirin (Experimental): All subjects in this arm (smokers (n=8) and non-smoking volunteers (n=8)) will receive 81 mg aspirin at approximately 8 am followed by 2000 mg acetaminophen at approximately 10 am during one crossover period (see "Crossover Period: Aspirin first" intervention). During the other crossover period, beginning after a 2 week washout, the order will be reversed and the subjects will receive 2000 mg acetaminophen at 8 am followed by 81 mg aspirin at 10 am (see "Crossover Period: Aspirin last" intervention). The occurrence of the two crossover periods will be randomized by order. Smokers and non-smokers will be matched for age and gender.
  Interventions: Drug: Aspirin First; Drug: Aspirin Last
- Phase 1b: Acetaminophen 1000 mg alone (Experimental): Eight male and non-pregnant female subjects who are healthy and non-smoking will be recruited. They will receive a daily oral dose of 1000 mg acetaminophen for six days each administered at 8 AM (see "Acetaminophen 1000 mg/d" intervention). Study assessments will be performed on day 1 and on day 6. This is not a crossover design. Just one treatment period.
  Interventions: Drug: Acetaminophen 1000 mg/d
- Phase 2: Acetaminophen vs. Ibuprofen (Experimental): Eight male and non-pregnant female subjects who are healthy and non-smoking will be recruited. In one period of this crossover study acetaminophen (1000 mg p.o.) will be administered orally at 8 AM, 2 PM, 8 PM and 2 AM for 3 days (see "Crossover Period: Acetaminophen 4000 mg/d" intervention). The last dose will be administered on day four at 8 AM In the other crossover period, after a washout period of at least 14 days, the subjects will receive ibuprofen (200 mg) orally at at 8 AM, 2 PM, 8 PM and 2 AM for 3 days (see "Crossover Period: Ibuprofen 800 mg/d" intervention). The last dose will be administered on day four at 8 AM Study assessments will be performed on day 1 and day 4 of each crossover period. The occurrence of the two crossover periods will be randomized by order.
  Interventions: Drug: Acetaminophen 4000 mg/d; Drug: Ibuprofen 800 mg/d

INTERVENTIONS:
Drug: Aspirin First — Crossover period Aspirin First: Subjects will receive 81 mg aspirin at approximately 8 am followed by acetaminophen at approximately 10 am.
  Arms: Phase 1a: Acetaminophen 1000mg / aspirin; Phase 1a: Acetaminophen 2000mg / aspirin
Drug: Aspirin Last — Crossover period Aspirin Last: Subjects will receive acetaminophen at approximately 8 am followed by 81 mg aspirin at approximately 10 am.
  Arms: Phase 1a: Acetaminophen 1000mg / aspirin; Phase 1a: Acetaminophen 2000mg / aspirin
Drug: Acetaminophen 1000 mg/d — Subjects will receive a daily oral dose of 1000 mg acetaminophen for six days each administered at 8 AM.
  Arms: Phase 1b: Acetaminophen 1000 mg alone
Drug: Acetaminophen 4000 mg/d — Crossover period Acetaminophen 4000 mg/d: Acetaminophen (1000 mg p.o.) orally at 8 AM, 2 PM, 8 PM and 2 AM for 3 days. The last dose will be administered on day four at 8 AM.
  Arms: Phase 2: Acetaminophen vs. Ibuprofen
Drug: Ibuprofen 800 mg/d — Crossover period Ibuprofen 800 mg/d: Ibuprofen (200 mg) orally at at 8 AM, 2 PM, 8 PM and 2 AM for 3 days. The last dose will be administered on day four at 8 AM.
  Arms: Phase 2: Acetaminophen vs. Ibuprofen

SUMMARY:
This research study investigates whether the ability of aspirin to reduce the risk of heart attacks may be diminished by the administration of acetaminophen. Patients who have heart disease are often prescribed aspirin because of its unique ability to permanently prevent platelets from aggregating and forming a blood clot. Such blood clots cause heart attacks when they form in a blood vessel that supplies the heart with oxygen rich blood. Some of these same patients also take acetaminophen everyday for relief from arthritis pain. Higher doses of acetaminophen may also have the ability to prevent the platelets from clotting, however only temporarily. Therefore, this study evaluates whether the timing of the administration of acetaminophen (before or after aspirin) interferes with the permanent blood clotting effects of aspirin.

The primary hypothesis is that acetaminophen given two hours before aspirin will antagonize the effects of aspirin, while reversing the order of administration will not.

DETAILED DESCRIPTION:
Acetaminophen has antipyretic and moderate analgesic properties, but largely lacks anti-inflammatory activity. While its mechanism of action is not entirely understood, it is probably both an isoform nonspecific and partial cyclooxygenase (COX) inhibitor in humans at doses commonly taken for mild pain and pyrexia, such as 1000 mg. Although no inhibition of platelet aggregation is observed at this dosage, platelet thromboxane formation by COX is depressed by roughly 40%. Epidemiological studies suggest that at higher doses, 2000 mg and above, acetaminophen exhibits a gastrointestinal adverse effect profile indistinguishable from traditional, nonspecific NSAIDs. Thus, it is possible that maximal COX inhibition is achieved at higher doses. Interestingly, complete COX inhibition by non-selective COX inhibitors has the potential to antagonize the irreversible platelet inhibition induced by aspirin. In contrast to reversible inhibitors, aspirin acts by acetylation of a serine residue in the substrate binding channel of COX. For example, ibuprofen, a reversible and non-selective COX inhibitor, is thought to prevent aspirin from gaining access to this target site. This study investigates, whether COX inhibition by acetaminophen is dose dependent in humans and whether acetaminophen interacts with the irreversible COX inhibition by low dose aspirin. It addresses the dose-related effect of acetaminophen on COX activity and assesses potential pharmacological interactions with low dose aspirin in normal healthy volunteers. The primary hypothesis is that administrating acetaminophen before aspirin would antagonize the irreversible effects of aspirin, as assessed by the measurement of serum thromboxane B2 24 hrs after the administration of the first study drug on day 6 of combination therapy.

The second aim will determine the effects of acetaminophen on oxidant stress and cyclooxygenase activity in patients who smoke. While the structural interaction of acetaminophen with COX is unknown, it may inactivate the enzyme by a molecular mechanism different from other NSAIDs. Thus, acetaminophen, which is a good reducing agent, might act to reduce COX from its active, oxidized form. When uninhibited, the peroxidase component of this bifunctional enzyme oxidizes its catalytic center to generate a tyrosyl radical that is required for its activity. Indeed, some reducing agents have the capacity to prevent COX activation in vitro. If reduction were the basis for COX inhibition by acetaminophen in vivo, it would be expected to be less pronounced under conditions of high peroxide tone, as occurs in inflammation. Indeed, acetaminophen, which is a phenol derivative, may act as a free radical scavenging antioxidant like other phenolic compounds, such as vitamin E and has been shown to alleviate oxidative damage in model systems. This study explores the potential antioxidant effect of acetaminophen in smokers. Such individuals represent a human model of oxidant stress. Novel approaches to the quantitative assessment of free radical induced damage to lipids are applied, which are elevated in smokers. Additionally, it is determined whether COX inhibition by acetaminophen is conditioned by oxidant tone in vivo.

The third aim, will compare the degree of COX inhibition by acetaminophen with that of a thoroughly characterized nonselective COX inhibitor, ibuprofen.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 - 55
* Subjects recruited for the "non-smoker group" must be in good health as based on medical history, physical examination, vital signs, and laboratory tests.
* Subjects recruited for the "smokers group" will be chronic smokers of at least 4 years duration, but no longer than 20 years duration, who smoke 11-20 cigarettes per day. Smokers must be otherwise healthy as described above.
* Female subjects of child bearing potential must be using a medically acceptable method of contraception (oral contraception, depo-provera injection, intrauterine device, condom with spermicide, diaphragm, cervical cap, progestin implant, abstinence, tubal ligation, oophorectomy, TAH) throughout the entire study period. All female subjects must consent to a urine pregnancy test at screening and just prior to the start of each treatment phase of the study, which must be negative at all time points.
* Subjects must be within 30% of their ideal body weight.

Exclusion Criteria:

* Female subjects who are pregnant or nursing a child.
* Subjects, who have received an experimental drug, used an experimental medical device within 30 days prior to screening, or who gave a blood donation of ≥ one pint within 8 weeks prior to screening.
* Subjects with any coagulation, bleeding or blood disorders.
* Subjects who are sensitive or allergic to acetaminophen and/or aspirin, as well as any of their components.
* Subjects with documented history of any gastrointestinal disorders, including bleeding ulcers.
* Subjects with any evidence of cancer.
* Subjects with a history of heart disease, including myocardial infarction, angina, coronary artery disease, any evidence of coronary artery stenosis, arrhythmias, heart failure, having had a coronary intervention or significant irregularities in the EKG.
* Subjects with history of peripheral artery disease (claudication, bypass surgery or stent placement in extremity.)
* Subjects with a history of stroke or transitory ischemic attacks.
* Subjects with renal, hepatic, respiratory, endocrine, metabolic, hematopoietic or neurological disorder.
* Subjects with a history of liver disease or abnormal liver function tests (>2x upper limit normal).
* Subjects with any abnormal laboratory value or physical finding that according to the investigator may interfere with interpretation of the study results, be indicative of an underlying disease state, or compromise the safety of a potential subject.
* Subjects who have had a history of drug or alcohol abuse within the last 6 months.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2004-06-02 (Actual); Primary Completion 2012-01-24 (Actual); Study Completion 2012-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Garret A. FitzGerald, MD, Principal Investigator — University of Pennsylvania, Institute for Translationals Medicine and Therapeutics; Susanne Fries, MD, Principal Investigator — University of Pennsylvania, Institute for Translationals Medicine and Therapeutics; Tilo Grosser, MD, Principal Investigator — University of Pennsylvania, Institute for Translationals Medicine and Therapeutics
Locations (1):
- Hospital of The University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Institute for Translational Medicine and Therapeutics, University of Pennsylvania — http://www.itmat.upenn.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase 1a: 16 evaluable healthy individuals and 16 evaluable apparently healthy chronic smokers. Crossover design.
  Phase 1b: 8 evaluable healthy and non-smoking subjects. No crossover.
  Phase 2: 8 evaluable healthy and non-smoking subjects. Crossover design.
  Enrollment from 6/2/2004 to 8/14/2007
Groups:
- Phase 1a: Aspirin 81 mg / Acetaminophen 1000 mg Sequence 1: All subjects in this arm of the study termed "Phase 1a" (smokers (n=8) and non-smokers (n=8) will receive 81 mg aspirin at 8 am followed by 1000 mg acetaminophen at 10 am each day, for six days during the first crossover period ("Aspirin first"). During the second crossover period, beginning after a 2 week washout, the order will be reversed and the subjects will receive 1000 mg acetaminophen at 8 am followed by 81 mg aspirin at 10 am each day, for six days ("Aspirin last"). The occurrence of the two crossover periods (interventions) will be randomized by order. Smokers and non-smokers will be matched for age and gender.
- Phase 1a: Aspirin 81 mg / Acetaminophen 1000 mg Sequence 2: All subjects in this arm of the study termed "Phase 1a" (smokers (n=8) and non-smokers (n=8) will receive 1000 mg acetaminophen at 8 am followed by 81 mg aspirin at 10 am each day, for six days during the first crossover period ("Aspirin last"). During the second crossover period, beginning after a 2 week washout, the order will be reversed and the subjects will receive 81 mg aspirin at 8 am followed by 1000 mg acetaminophen at 10 am each day, for six days ("Aspirin first"). The occurrence of the two crossover periods (interventions) will be randomized by order. Smokers and non-smokers will be matched for age and gender.
- Phase 1a: Aspirin 81 mg / Acetaminophen 2000 mg Sequence 1: All subjects in this arm of the study termed "Phase 1a" (smokers (n=8) and non-smokers (n=8) will receive 81 mg aspirin at 8 am followed by 2000 mg acetaminophen at 10 am each day, for six days during the first crossover period ("Aspirin first"). During the second crossover period, beginning after a 2 week washout, the order will be reversed and the subjects will receive 2000 mg acetaminophen at 8 am followed by 81 mg aspirin at 10 am each day, for six days ("Aspirin last"). The occurrence of the two crossover periods (interventions) will be randomized by order. Smokers and non-smokers will be matched for age and gender.
- Phase 1a: Aspirin 81 mg / Acetaminophen 2000 mg Sequence 2: All subjects in this arm of the study termed "Phase 1a" (smokers (n=8) and non-smokers (n=8) will receive 2000 mg acetaminophen at 8 am followed by 81 mg aspirin at 10 am each day, for six days during the first crossover period ("Aspirin last"). During the second crossover period, beginning after a 2 week washout, the order will be reversed and the subjects will receive 81 mg aspirin at 8 am followed by 2000 mg acetaminophen at 10 am each day, for six days ("Aspirin first"). The occurrence of the two crossover periods (interventions) will be randomized by order. Smokers and non-smokers will be matched for age and gender.
- Phase 1b: Acetaminophen 1000mg Alone: 4 Days: Eight healthy, non-smoking subjects will receive a daily oral dose of 1000 mg acetaminophen for six days each administered at 8 AM. Study assessments will be performed on day 1 and on day 6.
  Phase 1b is not a crossover design. Phase 1b will end after the first treatment period, which will be identical for all subjects.
- Phase 2: Acetaminophen 4000 mg/d / Ibuprofen 800 mg/d: In the first period of this arm of the crossover study termed "Phase 2", healthy non-smoking subjects will be administered acetaminophen (1000 mg) orally at 8 AM, 2 PM, 8 PM and 2 AM (4000 mg/d) for 3 days. The last dose will be administered on day four at 8 AM In the other crossover period, after a washout period of at least 14 days, the subjects will receive ibuprofen (200 mg) orally at 8 AM, 2 PM, 8 PM and 2 AM (800 mg/d) for 3 days. The last dose will be administered on day four at 8 AM. The treatment periods will be randomized by order.
- Phase 2: Ibuprofen 800 mg/d / Acetaminophen 4000 mg/d: In the first period of this arm of the crossover study termed "Phase 2", healthy non-smoking subjects will be administered ibuprofen (200 mg) orally at 8 AM, 2 PM, 8 PM and 2 AM (800 mg/d) for 3 days. The last dose will be administered on day four at 8 AM In the other crossover period, after a washout period of at least 14 days, the subjects will receive acetaminophen (1000 mg) orally at 8 AM, 2 PM, 8 PM and 2 AM (4000 mg/d) for 3 days. The last dose will be administered on day four at 8 AM. The treatment periods will be randomized by order.
Period: Crossover Period 1
Arm/Group | Phase 1a: Aspirin 81 mg / Acetaminophen 1000 mg Sequence 1 | Phase 1a: Aspirin 81 mg / Acetaminophen 1000 mg Sequence 2 | Phase 1a: Aspirin 81 mg / Acetaminophen 2000 mg Sequence 1 | Phase 1a: Aspirin 81 mg / Acetaminophen 2000 mg Sequence 2 | Phase 1b: Acetaminophen 1000mg Alone: 4 Days | Phase 2: Acetaminophen 4000 mg/d / Ibuprofen 800 mg/d | Phase 2: Ibuprofen 800 mg/d / Acetaminophen 4000 mg/d
Started | 9 | 9 | 10 | 9 | 8 | 5 | 5
Completed | 8 | 9 | 10 | 9 | 8 (Phase 1b had only one treatment period and no crossover. Phase 1b ended here.) | 4 | 5
Not Completed | 1 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 1 | 0
Period: Washout (>/= 14 Days)
Arm/Group | Phase 1a: Aspirin 81 mg / Acetaminophen 1000 mg Sequence 1 | Phase 1a: Aspirin 81 mg / Acetaminophen 1000 mg Sequence 2 | Phase 1a: Aspirin 81 mg / Acetaminophen 2000 mg Sequence 1 | Phase 1a: Aspirin 81 mg / Acetaminophen 2000 mg Sequence 2 | Phase 1b: Acetaminophen 1000mg Alone: 4 Days | Phase 2: Acetaminophen 4000 mg/d / Ibuprofen 800 mg/d | Phase 2: Ibuprofen 800 mg/d / Acetaminophen 4000 mg/d
Started | 8 | 9 | 10 | 9 | 0 (Phase 1b had only one treatment period and no crossover.) | 4 | 5
Completed | 8 | 9 | 10 | 9 | 0 (Phase 1b had only one treatment period and no crossover.) | 4 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Crossover Period 2
Arm/Group | Phase 1a: Aspirin 81 mg / Acetaminophen 1000 mg Sequence 1 | Phase 1a: Aspirin 81 mg / Acetaminophen 1000 mg Sequence 2 | Phase 1a: Aspirin 81 mg / Acetaminophen 2000 mg Sequence 1 | Phase 1a: Aspirin 81 mg / Acetaminophen 2000 mg Sequence 2 | Phase 1b: Acetaminophen 1000mg Alone: 4 Days | Phase 2: Acetaminophen 4000 mg/d / Ibuprofen 800 mg/d | Phase 2: Ibuprofen 800 mg/d / Acetaminophen 4000 mg/d
Started | 8 | 9 | 10 | 9 | 0 (Phase 1b had only one treatment period and no crossover.) | 4 | 5
Completed | 8 | 8 | 8 | 8 | 0 (Phase 1b had only one treatment period and no crossover.) | 4 | 4
Not Completed | 0 | 1 | 2 | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Phase 1a: Acetaminophen 1000mg / Aspirin: All subjects in this arm (smokers (n=8) and non-smokers (n=8) will receive 81 mg aspirin at approximately 8 am followed by 1000 mg acetaminophen at approximately 10 am during one treatment phase (see "Aspirin first" intervention). During the other treatment phase, beginning after a 2 week washout, the order will be reversed and the subjects will receive 1000 mg acetaminophen at 8 am followed by 81 mg aspirin at 10 am (see "Aspirin last" intervention). The occurrence of the two study phases (interventions) will be randomized by order. Smokers and non-smokers will be matched for age and gender.
  Aspirin first: Subjects will receive 81 mg aspirin at approximately 8 am followed by 1000 or 2000 mg acetaminophen at approximately 10 am during this intervention phase.
  Aspirin last: Subjects will receive 1000 or 2000 mg acetaminophen at approximately 8am followed by 81 mg aspirin at approximately 10 am during this intervention phase.
- Phase 1a: Acetaminophen 2000mg / Aspirin: All subjects in this arm (smokers (n=8) and non-smoking volunteers (n=8)) will receive 81 mg aspirin at approximately 8 am followed by 2000 mg acetaminophen at approximately 10 am during one treatment phase (see "Aspirin first" intervention). During the other treatment phase, beginning after a 2 week washout, the order will be reversed and the subjects will receive 2000 mg acetaminophen at 8 am followed by 81 mg aspirin at 10 am (see "Aspirin last" intervention). The occurrence of the two study phases (interventions) will be randomized by order. Smokers and non-smokers will be matched for age and gender.
  Aspirin first: Subjects will receive 81 mg aspirin at approximately 8 am followed by 1000 or 2000 mg acetaminophen at approximately 10 am during this intervention phase.
  Aspirin last: Subjects will receive 1000 or 2000 mg acetaminophen at approximately 8am followed by 81 mg aspirin at approximately 10 am during this intervention phase.
- Phase 1b: Acetaminophen 1000 mg Alone: Eight male and non-pregnant female subjects who are healthy and non-smoking will be recruited. They will receive a daily oral dose of 1000 mg acetaminophen for six days each administered at 8 AM (see "Acetaminophen 1000 mg/d" intervention). Study assessments will be performed on day 1 and on day 6.
  Acetaminophen 1000 mg/d: They will receive a daily oral dose of 1000 mg acetaminophen for six days each administered at 8 AM.
- Phase 2: Acetaminophen vs. Ibuprofen: Eight male and non-pregnant female subjects who are healthy and non-smoking will be recruited. In one treatment period of this cross-over study acetaminophen (1000 mg p.o.) will be administered orally at 8 AM, 2 PM, 8 PM and 2 AM for 3 days (see "Acetaminophen 4000 mg/d" intervention). The last dose will be administered on day four at 8 AM In the other treatment period, after a washout period of at least 14 days, the subjects will receive ibuprofen (200 mg) orally at at 8 AM, 2 PM, 8 PM and 2 AM for 3 days (see "Ibuprofen 800 mg/d" intervention). The last dose will be administered on day four at 8 AM.
  Acetaminophen 4000 mg/d: Acetaminophen (1000 mg p.o.) orally at 8 AM, 2 PM, 8 PM and 2 AM for 3 days. The last dose will be administered on day four at 8 AM.
  Ibuprofen 800 mg/d: Ibuprofen (200 mg) orally at at 8 AM, 2 PM, 8 PM and 2 AM for 3 days. The last dose will be administered on day four at 8 AM.
- Total: Total of all reporting groups
Arm/Group | Phase 1a: Acetaminophen 1000mg / Aspirin | Phase 1a: Acetaminophen 2000mg / Aspirin | Phase 1b: Acetaminophen 1000 mg Alone | Phase 2: Acetaminophen vs. Ibuprofen | Total
Number analyzed (Participants) | 16 | 16 | 8 | 8 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 16 | 8 | 8 | 48
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.3 (11.4) | 37.6 (11.2) | 31.8 (7.1) | 30.9 (8.3) | 33.9 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 3 | 4 | 23
  Male | 8 | 8 | 5 | 4 | 25
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 8 | 8 | 48

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Serum Thromboxane B2
Description: Thromboxan B2 is a stable metabolite of thromboxane A2. Thromboxane B2 formation during clotting of whole blood (37 degrees Celsius, 1 hour) is reflective of the capacity of platelets to form thromboxane A2. Serum Thromboxane B2 was measured by radio-immuno assay. The quantity of interest was percent change from start (8:00 am on day 1) to finish (8:00 am on last day) of each crossover period in serum thromboxane B2. This was calculated as: 100%*(value at start of period minus value at end of period)/value at start of period.
Time Frame: 7 days (Phase 1a and 1b), 4 days (Phase 2)
Measure: Mean (Standard Deviation); unit: Percent inhibition of baseline
Groups:
- Phase 1a: Acetaminophen 1000 mg / Aspirin First: 81 mg aspirin at 8 am followed by 1000 mg acetaminophen at 10 am.
- Phase 1a: Acetaminophen 1000 mg / Aspirin Last: 1000 mg acetaminophen at 8am followed by 81 mg aspirin at 10 am.
- Phase 1a: Acetaminophen 2000 mg / Aspirin First: 81 mg aspirin at 8 am followed by 2000 mg acetaminophen at 10 am.
- Phase 1a: Acetaminophen 2000 mg / Aspirin Last: 2000 mg acetaminophen at 8am followed by 81 mg aspirin at 10 am.
- Phase 1b: Acetaminophen 1000 mg/d: Eight male and non-pregnant female subjects who are healthy and non-smoking will be recruited. They will receive a daily oral dose of 1000 mg acetaminophen for six days each administered at 8 AM (see "Acetaminophen 1000 mg/d" intervention). Study assessments will be performed on day 1 and on day 6.
  Acetaminophen 1000 mg/d: They will receive a daily oral dose of 1000 mg acetaminophen for six days each administered at 8 AM.
- Phase 2: Acetaminophen 4000 mg/d: Acetaminophen (1000 mg p.o.) orally at 8 AM, 2 PM, 8 PM and 2 AM for 3 days. Last dose on day four at 8 AM.
- Phase 2: Ibuprofen 800 mg/d: Ibuprofen (200 mg) orally at at 8 AM, 2 PM, 8 PM and 2 AM for 3 days. Last dose on day four at 8 AM.
Arm/Group | Phase 1a: Acetaminophen 1000 mg / Aspirin First | Phase 1a: Acetaminophen 1000 mg / Aspirin Last | Phase 1a: Acetaminophen 2000 mg / Aspirin First | Phase 1a: Acetaminophen 2000 mg / Aspirin Last | Phase 1b: Acetaminophen 1000 mg/d | Phase 2: Acetaminophen 4000 mg/d | Phase 2: Ibuprofen 800 mg/d
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 8 | 8 | 8
Percent inhibition of baseline | 97.0 (4.7) | 97.4 (3.6) | 98.3 (1.0) | 96.7 (2.6) | -6.5 (59.7) | 21.9 (19.7) | 62.6 (32.2)
Statistical Analysis 1: Comparison: Phase 1a: Acetaminophen 1000 mg / Aspirin First vs Phase 1a: Acetaminophen 1000 mg / Aspirin Last vs Phase 1a: Acetaminophen 2000 mg / Aspirin First vs Phase 1a: Acetaminophen 2000 mg / Aspirin Last; The primary hypothesis is that acetaminophen given two hours before aspirin will antagonize the effects of aspirin, while reversing the order of administration will not. Percent change from start (8:00 am on day 1) to finish (8:00 am on day 7) of period in serum thromboxane B2 for each order of drug administration will be primary endpoint of interest; Test type: Superiority — An analysis of variance, appropriate for a three factor experiment with cohort and dose as non-repeated factors and repeated measure order arranged in a two period cross-over design, was performed; p > 0.05, ANOVA

2. Secondary Outcome: Percent Change in Arachidonic Acid Induced Platelet Aggregation
Description: Platelet aggregation was induced by 500 micro molar arachidonic acid using a Chronolog aggregometer. The quantity of interest was percent change from start (8:00 am on day 1) to finish (8:00 am on last day) of each crossover period in platelet aggregation. This was calculated as: 100%*(value at start of period minus value at end of period)/value at start of period.
Time Frame: 7 days (only Phase 1a)
Measure: Mean (Standard Deviation); unit: Percent inhibition of baseline
Arm/Group | Phase 1a: Acetaminophen 1000 mg / Aspirin First | Phase 1a: Acetaminophen 1000 mg / Aspirin Last | Phase 1a: Acetaminophen 2000 mg / Aspirin First | Phase 1a: Acetaminophen 2000 mg / Aspirin Last
Number analyzed (Participants) | 16 | 16 | 16 | 16
Percent inhibition of baseline | 93 (6) | 93 (6) | 95 (4) | 90 (16)
Statistical Analysis 1: Comparison: Phase 1a: Acetaminophen 1000 mg / Aspirin First vs Phase 1a: Acetaminophen 1000 mg / Aspirin Last vs Phase 1a: Acetaminophen 2000 mg / Aspirin First vs Phase 1a: Acetaminophen 2000 mg / Aspirin Last; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p > 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: Phase 1a: Approximately 4 weeks (depending on the length of the washout period between treatment periods). Phase 1b: 4 days. Phase 2: Approximately 4 weeks (depending on the length of the washout period between treatment periods).
Arm/Group | Phase 1a: Acetaminophen 1000mg / Aspirin | Phase 1a: Acetaminophen 2000mg / Aspirin | Phase 1b: Acetaminophen 1000 mg Alone | Phase 2: Acetaminophen vs. Ibuprofen
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes